CLINICAL TRIAL: NCT01568944
Title: Peripheral Blood Dendritic Cells and Periodontitis
Brief Title: Role of Infected Blood Dendritic Cells in Heart Disease Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Christopher Cutler, Assoc. Dean Dental Medicine, Dept. Chair Periodontics, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R21DE020916 (NIH); Pro00000394 (Other: GHSU-HAC); R21DE020916 (NIH)
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Chronic Periodontitis
Keywords: periodontal; disease; dendritic; cells; antibiotics
MeSH Terms: conditions — Chronic Periodontitis; Disease | interventions — Anti-Bacterial Agents; Mouthwashes; chlorhexidine gluconate; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Antibiotic and Oral Rinse (Experimental): Each subject will received oral Amoxicillin/Amoxil/lansoprazole/Flagyl 250 mg of each three times a day for 8 days. Subjects will also rinse their mouths with 2 ounces of 0.12% chlorhexidine/peridex mouthrinse two times per day. Subjects will also receive mechanical debridement at the baseline visit. Intervention Amoxicillin/Amoxil/lansoprazol 500 mg/ Metronidazole/Flagyl 250 mg
  Interventions: Drug: Oral Antibiotic and Oral Rinse; Procedure: Standard Treatment
- Standard Treatment (Other): Subjects assigned to standard treatment will receive full mouth scaling and root planing using hand instrumentation (curettes) and ultrasonic scalers
  Interventions: Procedure: Standard Treatment

INTERVENTIONS:
Drug: Oral Antibiotic and Oral Rinse — PO Amoxicillin in 500 mg / Metronidazole 250 mg of each TID for 8 days plus 2 ounces of 0.12% chlorhexidine mouthrinse used BID
  Other Names: Peridex/Flagyl/Amoxil/lansoprazole
  Arms: Oral Antibiotic and Oral Rinse
Procedure: Standard Treatment — Full mouth scaling and root planing using hand instrumentation (curettes) and ultrasonic scalers
  Other Names: Scaling; Root planing

SUMMARY:
The investigators hypothesize that blood dendritic cells harbor pathogens from the oral cavity in chronic periodontitis and disseminate these pathogens to atherosclerotic plaques.

DETAILED DESCRIPTION:
To address this hypothesis, a clinical study in humans with moderate to severe chronic periodontitis has been designed. This is an interventional study involving scaling and root planing and two arms: 1. treatment with PO amoxocillin/metronidazole plus chlorhexidine oral rinse; 2. no antibiotics or oral rinse. It is expected that the antibiotics plus chlorhexidine will prevent the dendritic cell response to infection (bacteremia) elicited by scaling and root planing.

ELIGIBILITY:
Inclusion Criteria:

* generalized moderate to severe chronic periodontitis

Exclusion Criteria:

* diabetes
* antibiotics treatment within 3 months
* treatment with steroids, phenytoin, cyclosporin, coumadin
* presence of conditions requiring prophylactic antibiotics per AHA
* cancer, HIV, hepB, lupus, prediagnosed heart disease, renal disease
* smoker

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cutler, DDS, Principal Investigator — GHSU-College of Dental Medicine
Locations (1):
- GHSU-CDM Clinical Research Center, Augusta, Georgia, United States

REFERENCES:
- [Background] Zeituni AE, McCaig W, Scisci E, Thanassi DG, Cutler CW. The native 67-kilodalton minor fimbria of Porphyromonas gingivalis is a novel glycoprotein with DC-SIGN-targeting motifs. J Bacteriol. 2010 Aug;192(16):4103-10. doi: 10.1128/JB.00275-10. Epub 2010 Jun 18. PMID 20562309
- [Background] Zeituni AE, Carrion J, Cutler CW. Porphyromonas gingivalis-dendritic cell interactions: consequences for coronary artery disease. J Oral Microbiol. 2010 Dec 21;2. doi: 10.3402/jom.v2i0.5782. PMID 21523219

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Started | 8 | 10
Completed | 8 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (4) | 48 (5) | 46 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Blood Dendritic Cells From Baseline
Description: The frequency of blood dendritic cells, i.e. % CCR6+CD1a+ DCs by flow cytometry 30 days after treatment with 7 day regimen of antibiotics, mouthrinse therapy and scaling and root planing (SRP) will be compared to those who did not receive the antibiotics, but did receive mouthrinse and scaling and root planing (SRP)
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: % MFI
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Number analyzed (Participants) | 8 | 10
% MFI | 12 (4) | 14 (2)

2. Secondary Outcome: Probing Attachment Levels
Description: Probing attachment levels (distance from the cemento-enamel junction to the base of the periodontal pocket in mm at 6 sites p[er tooth) will be monitored after 30 days
Time Frame: 30 days
Population: The number of teeth
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: tooth sites
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Number analyzed (Participants) | 8 | 10
Number analyzed (tooth sites) | 32 | 32
mm | 4.2 (6) | 4.6 (4)

3. Secondary Outcome: Serum Cytokine Response
Description: serum CCL20 in pg/ml by ELISA will be measured after 30 days
Time Frame: 30 days
Population: CCL20 in pg/ml of serum will be measured by ELISA
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Number analyzed (Participants) | 8 | 10
pg/ml | 22 (5) | 32 (5)

4. Secondary Outcome: Probing Depths
Description: Probing depths (distance from the free gingival margin to the base of the pocket in mm at six sites per tooth) will be monitored after 30 days
Time Frame: 30 days
Population: Probing depths in mm at 192 sites per patient
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: sites per mouth
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Number analyzed (Participants) | 8 | 10
Number analyzed (sites per mouth) | 192 | 192
mm | 4.2 (3) | 4.7 (4)

5. Secondary Outcome: Plaque Index
Description: Plaque index of Silness and Loe will be monitored at buccal and lingual surfaces of all teeth after 30 days:
  0 no visible microbial plaque
  1. thin film of visible microbial plaque in sulcus
  2. moderate accumulation of plaque in sulcus
  3. large amount of plaque in sulcus or along free gingival margin
Time Frame: 30 days
Population: plaque index at 64 sites per mouth will be measured
Measure: Median (90% Confidence Interval); unit: pI index
Units Other Than Participants: sites per mouth
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Number analyzed (Participants) | 8 | 10
Number analyzed (sites per mouth) | 64 | 64
pI index | 2 [0 to 3] | 3 [1 to 3]

6. Secondary Outcome: Gingival Index
Description: Gingival index of Loe and Silness on facial, lingual and mesial surfaces of all teeth will be monitored after 30 days:
  0 Normal, no inflammation
  1. Mild inflammation, slight color change and edema, no bleeding
  2. Moderate inflammation, redness, edema, bleeds on probing
  3. Severe inflammation, marked redness and edema ulceration, spontaneous bleeding
Time Frame: 30 days
Population: gingival index at 3 sites per tooth
Measure: Median (90% Confidence Interval); unit: GI
Units Other Than Participants: 3 sites per tooth
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
Number analyzed (Participants) | 8 | 10
Number analyzed (3 sites per tooth) | 96 | 96
GI | 2 [1 to 3] | 3 [2 to 4]

ADVERSE EVENTS:
Time Frame: 30 days
Description: The antibiotic protocol is reported to induce gastric upset, diarrhea and/or vaginal candidiasis in some subjects. All subjects were asked if they had any of these symptoms and none were reported
Arm/Group | Oral Antibiotic and Oral Rinse | Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No